CLINICAL TRIAL: NCT06030492
Title: Efficacy of Hydrogen Peroxide ( H2O2) in Controlling Placental Site Bleeding in Caesarian Delivery for Placenta Previa / Accreta Spectrum ( PAS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassiony Dabian, lecturer of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-467-2023
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrogen peroxide group (Experimental): hydrogen peroxide group Irrigation of the placental bed with 100 ml 3% hydrogen peroxide , followed by packing with a towel highly soaked hydrogen peroxide solution (Pozitif Kimya, İstanbul, Turkey) , freshly prepared by a 50% dilution with a normal saline solution.(
  Interventions: Drug: packing placental site with hydrogen peroxide soaked towels
- normal Saline solution (Placebo Comparator): Packing the placental bed with a towel soaked with normal Saline solution
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: packing placental site with hydrogen peroxide soaked towels — Skin is incised either midline or Pfannenstiel incision according to clinical situation , bladder dissection will be done , uterus will be incised by transverse lower segment incision , followed by delivery of the baby.
  Uterine massage , ecbolics & a trial for delivery of the placenta will be done Irrigation of the placental bed with 100 ml 3% hydrogen peroxide , followed by packing with a towel highly soaked hydrogen peroxide solution (Pozitif Kimya, İstanbul, Turkey) , freshly prepared by a 50% dilution with a normal saline solution
  Arms: hydrogen peroxide group
Drug: normal Saline — Skin is incised either midline or Pfannenstiel incision according to clinical situation , bladder dissection will be done , uterus will be incised by transverse lower segment incision , followed by delivery of the baby.
  Uterine massage , ecbolics & a trial for delivery of the placenta will be done.
  Packing the placental bed with a towel soaked with normal Saline solution
  Arms: normal Saline solution

SUMMARY:
Placenta accreta spectrum (PAS), encompassing the terms placenta accreta, increta, and percreta; abnormally invasive placenta; morbidly adherent placenta; and invasive placentation, is a leading cause of life-threatening obstetric haemorrage (1) . Currently, more than 90% of women diagnosed with PAS also have a placenta praevia (2), and the combination of both conditions leads to high maternal morbidity and mortality due to massive haemorrhage at the time of birth . Maternal mortality of placenta praevia with percreta has been reported to be as high as 7% of cases .

Hydrogen peroxide is well-known for its antimicrobial and antiseptic properties. It is used to clean surgical cuts for better localization of bleeding focus in surgery and orthopedics and burn excisions to induce hemostasis . Topical application of hydrogen peroxide was proven to induce hemostasis and reduce operative time in both tonsillectomy and adenoidectomy .

DETAILED DESCRIPTION:
* Population of study: A total of 84 pregnant patients with placenta previa / Accreta spectrum.
* Study location: Obstetrics and Gynecology Kasr Al-Ainy Hospital , Faculty of Medicine , Cairo University.

The aim of the study is to evaluate the efficacy of hydrogen peroxide for controlling bleeding from placental bed in caesarian section for placenta previa/ Accreta spectrum (PAS).

• This is a randomized controlled trial including a total number of 84 patients representing study group , randomized in 2 equal groups , using computer generated randomization sheet on (Medcalc ®) .

Group A : hydrogen peroxide group (n=42)

Group B : control group (normal Saline solution) (n=42) .

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-40 years
* BMI < 35 kg/m2
* Pregnant patients with placenta previa .
* Placenta accrete FIGO grade 1 .
* Vitally stable .
* Candidate for conservative management.
* No major intra-operative bleeding.

Exclusion Criteria:

* Vitally unstable .
* Massive pre- or intra-operative bleeding.
* Medical disorders ( e.g. : hypertension , cardiac …. )
* Placenta accrete , FIGO grades 2 or 3 .
* Not indicated for conservative management.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
control of intra-operative bleeding from placental bed | 3 minutes after application of topical drug , identified as arrest of bleeding or minimal oozing from placental bed with good general condition & no hemoglobin drop
  control of intra-operative bleeding from placental bed

SECONDARY OUTCOMES:
Estimated intraoperative blood loss | from begining to end of surgery
  Estimated intraoperative blood loss by towel saturarion , amount of blood in suction , and pre& postoperative hemoglobin and hematocrite
Need for hemostatic sutures , uterine artery ligation , internal iliac artery ligation , hysterectomy | 3 minutes after topical application , if bleeding continued
  Need for hemostatic sutures , uterine artery ligation , internal iliac artery ligation , hysterectomy
immediate maternal complications ( postpartum haemorrage , DIC , hysterectomy , maternal mortality , ICU admission , …) | within 1st 24 hours postoperative
  immediate maternal complications ( postpartum haemorrage , DIC , hysterectomy , maternal mortality , ICU admission , …)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy outpatient infertility clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sheiner E, Sarid L, Levy A, Seidman DS, Hallak M. Obstetric risk factors and outcome of pregnancies complicated with early postpartum hemorrhage: a population-based study. J Matern Fetal Neonatal Med. 2005 Sep;18(3):149-54. doi: 10.1080/14767050500170088. PMID 16272036
- [Background] Jauniaux E, Bhide A, Kennedy A, Woodward P, Hubinont C, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Prenatal diagnosis and screening. Int J Gynaecol Obstet. 2018 Mar;140(3):274-280. doi: 10.1002/ijgo.12408. No abstract available. PMID 29405319
- [Background] Wasserbauer S, Perez-Meza D, Chao R. Hydrogen peroxide and wound healing: a theoretical and practical review for hair transplant surgeons. Dermatol Surg. 2008 Jun;34(6):745-50. doi: 10.1111/j.1524-4725.2008.34141.x. Epub 2008 Mar 3. PMID 18318724